CLINICAL TRIAL: NCT01604031
Title: Treatment of B-CLL With Autologous IL2 and CD40 Ligand-Expressing Tumor Cells + Lenalidomide
Acronym: TAIL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Martha Mims, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-30087 TAIL
Record Dates: First submitted 2012-05-04; First posted 2012-05-23 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: B-cell Chronic Lymphocytic Leukemia
Keywords: B-CLL; vaccine; Lenalidomide; CTL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- B-CLL vaccine (Experimental): Patients will receive doses of vaccine at 2 week intervals for 5 doses and at 4 week intervals for doses 6-16. The injection will be performed subcutaneously in the deltoid region of the upper arm.
  Interventions: Biological: B-CLL Vaccine; Drug: Lenalidomide

INTERVENTIONS:
Biological: B-CLL Vaccine — Patients will receive a fixed dose (2X10^7) of IL-2 secreting B-cells together with (2X10^7) of hCD40L expressing B-cells. Patients will receive doses of vaccine at 2 week intervals for 5 doses. Barring adverse events, an additional 11 doses of vaccine will be given, at 4 weekly intervals beginning on week 12 for a total period of one year or 16 vaccinations in total.
Drug: Lenalidomide — Subjects will begin lenalidomide 5 mg orally daily on day zero and will continue daily dosing until week 60 (4 weeks after the final dose of vaccine).
  Other Names: Revlimid

SUMMARY:
This is a research study to determine the safety and effectiveness of using special cells that may make the subject's immune system fight their chronic lymphocytic leukemia (CLL) in combination with a drug called Lenalidomide.

To do this, the investigators will put a special gene into cancer cells that have been taken from the subject. This will be done in the laboratory. This gene will make the cells produce interleukin 2 (IL-2), which is a natural substance that may help the subject's immune system kill cancer cells. Additionally, the investigators will stimulate the cancer cells with normal embryonic fibroblasts (cells that develop into normal connective tissues in the body) so that they will make another natural protein called CD40 ligand (CD40L). Some of these cells will then be put back into the subject's body with the goal that they will act like a vaccine and stimulate the immune system to attack the CLL cells.

The investigators have already conducted a study similar to this in other subjects with CLL. In those subjects the investigators saw some changes in the subject's immune system that might indicate that the modified cells were helping their immune system fight the cancer. However, in most of the subjects this change in the immune system went away after the injections were stopped. The investigators think that this may be due to a high level of cells called T regulatory cells. T regulatory cells are part of the immune system and prevent excessive reactions from other cells in the body. Studies have shown that reducing T regulatory cells allows the body to fight the cancer for a longer period of time.

Recent studies have shown that using Lenalidomide helps the body reduce T regulatory cells. Using Lenalidomide along with the injections (shots) might help the body fight the cancer for a longer period of time. Lenalidomide is also called Revlimid.

In this study the investigators want to see if they can make the change in the immune system last longer by giving Lenalidomide before and at the same time as the vaccine. The investigators hope that this might produce a better response directed at the CLL cells. Subjects will receive injections for about a year

DETAILED DESCRIPTION:
Previously, some of the cancer cells were taken from the subject's body and separated in the laboratory and a specially produced human virus (adenovirus) that carries the IL-2 gene was put into the cells. Adenovirus is a common virus found in human respiratory systems. In its normal state, it can reproduce and cause a respiratory infection. Respiratory illnesses caused by adenovirus infections range from the common cold to pneumonia, croup and bronchitis. This adenovirus has been changed in the laboratory so that it is not likely to reproduce or cause an infection once it is in the body. The gene transfer method used in this study tries to add copies of the IL2 gene that increases the immune response against a tumor.

The rest of the cancer cells have been stimulated to express on their surface a substance called the human CD40L. These substances (IL-2 and CD40L), already naturally present in the body, are meant to help the immune system fight the cancer.

At the point that the doctor feels the subject should begin treatment on this protocol, the treatment will be as follows:

The subject will begin taking Allopurinol by mouth at 300 mg and will continue taking Allopurinol daily for 14 days. Allopurinol is also called Zyloprim and it will be taken to prevent tumor lysis syndrome. Tumor lysis syndrome can be a serious condition that occurs sometimes when cancer treatment is started. Tumor lysis syndrome can cause other medical problems.

Two days after Allopurinol was started, the subject will begin taking Lenalidomide. The Lenalidomide dose will be 5 mg taken by mouth daily. The subject should swallow the capsules whole with water at the same time each day and should not break, chew or open the capsules. Females of childbearing potential who are caring for the subject should not touch the lenalidomide capsules or bottles without gloves. If a dose of lenalidomide is missed, it should be taken as soon as possible on the same day. If it is missed for the entire day, it should not be made up. If more than the prescribed dose is taken of lenalidomide and the subject feels poorly, s/he should seek emergency medical care and tell the study staff right away. The subject will get 1 cycle of drug per month. A max of a 28-day supply of the drug will be provided at one time. If the subject has bad side effects the doctor may tell him/her not to take the lenalidomide for a short time period or may be removed from the study. Otherwise, the subject will continue daily dosing with Lenalidomide for approximately 1 year, until four weeks after the final vaccine.

Four weeks after the subject starts the Lenalidomide s/he will start to receive his/her vaccines. The vaccine will be injected under the skin (also called subcutaneously). Normally the subject will have the shots as an outpatient (no overnight stay in the hospital will be required). S/he will receive the first five (5) shots at 2 week intervals. S/he will then receive eleven (11) shots at 4 weekly intervals. In total, the subject may receive up to sixteen (16) shots over a period of one year. As with the Lenalidomide if the subject has bad side effects s/he may not receive his/her vaccines for a short period of time or may be removed from the study. Otherwise, the subject will receive the vaccines on the schedule as specified earlier in this paragraph. These shots must be given at Houston Methodist Hospital.

Following these injections, the doctor will follow the subject for 1 year after the last shot to see how the subject is doing.

TESTS DURING AND AFTER EXPERIMENTAL TREATMENT:

A complete history and physical examination is necessary before the subject can be enrolled in the study. A physical examination will also be performed each time s/he receives a shot of the modified cells. The place on the subject's body where s/he had received the shots will be examined during the physical exam.

Research Blood Samples:

Blood will be taken from a tube placed into the vein (IV). We will take blood samples at the following time points: at study entry, week 0 when the subject starts Lenalidomide, weeks 2, 4, 6, 8, 10 and 16 and then every 4 weeks until week 60. The last blood sample will be at one year after the last shot. We will do this to make sure that the Lenalidomide is working correctly and to study how the modified cells are working in the body.

The amount of blood that will be obtained each time is approximately 2-3 tablespoonfuls, which is considered to be a safe amount. If the subject has a central line (an IV line that has been placed in a large blood vessel that is meant to be used for long periods of time), the blood will be taken from it, so that extra "sticks" should not be needed. Additional office visits may be necessary to obtain this blood. The maximum total amount of blood to be collected from the subject is 40-60 tablespoons.

Other tests: If the subject is a woman who can get pregnant, she will have pregnancy counseling and urine tests as long as she is taking lenalidomide.

In order to participate in this study, the subject must register into and follow the requirements of the Revlimid REMS® program of Celgene Corporation (the company that supplies Lenalidomide). This program provides education and counseling on the risks of fetal exposure, blood clots and reduced blood counts that can occur when taking Lenalidomide. The subject will be required to receive counseling every 28 days during treatment with lenalidomide, follow the pregnancy testing and birth control requirements of the program that are appropriate for him/her and take telephone surveys regarding your compliance with the program. Participating in the Revlimid REMS® program is a study requirement.

ELIGIBILITY:
Inclusion Criteria:

ELIGIBILITY FOR BLAST COLLECTION (procurement):

* Patients with B-CLL (not in Richter's transformation) with measurable disease.
* Procurement consent signed and faxed to Research Coordinator
* HIV negative (can be pending at this time)

ELIGIBILITY FOR VACCINE AND LENALIDOMIDE ADMINISTRATION (protocol entry):

* Manipulated B-CLL cells available (at least 6 injections)
* Patients with B-CLL (not in Richter's transformation) with measurable disease
* Patients must have a life expectancy of at least 10 weeks.
* Patients must be less than 75 years old
* Patients must have ECOG performance status of 0-2.
* Patients must have recovered from the toxic effects of all prior chemotherapy before entering this study:
* Absolute neutrophil count (ANC) of greater than or equal to 500/microL
* Absolute lymphocyte count (ALC) greater than or equal 200/microL,
* Hemoglobin greater than or equal 8 g/dL
* Platelet count greater than or equal 50,000/microL.
* Patients must be willing to practice appropriate birth control methods during the study and for 28 days after their participation in the treatment portion of the study is concluded.
* Patients must have adequate liver function:
* Total bilirubin less than or equal to 1.5 mg/dl, SGOT less than or equal to 3 times normal
* Normal prothrombin time
* Patients must have adequate renal function (creatinine clearance greater than 50 ml/min).
* Patients provide informed consent.
* Patient must not have received treatment with other investigational agents within the last 4 weeks.
* All study participants (treatment) must be registered in the REMS® Program and be willing to comply with the requirements of REMS® .

Note: A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

EXCLUSION CRITERIA FOR VACCINE ADMINISTRATION (protocol entry):

* Infected at time of protocol entry, or receiving antibiotics (other than prophylactic trimethoprim sulfamethoxazole).
* Pregnant or lactating
* Suffering from an autoimmune disease (including refractory immune thrombocytopenia-ITP or refractory autoimmune hemolytic anemia-AIHA)
* Receiving immunosuppressive drugs.
* Received systemic steroids within 30 days of study enrollment
* Autologous hematopoietic stem cell transplant or fludarabine chemotherapy within 6 months of study enrollment
* History of allogeneic stem cell transplant
* Patients with congestive heart failure or significant arrhythmia
* Known hypersensitivity to thalidomide or lenalidomide.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Adverse Events after Lenalidomide with B-CLL cell vaccine | week 60
  To assess the safety of administration of lenalidomide combined with prolonged administration of CD40L expressing and IL-2 secreting B-CLL cells (B-CLL vaccine).
Changes in SP tumor cell population from pre-vaccine to four weeks post-vaccination | week 4
  To determine the effects of administration of lenalidomide combined with CD40L expressing and IL-2 secreting B-CLL cells on overall disease burden and on the side population of tumor cells.
Changes in SP tumor cell population from pre-vaccine to eight weeks post vaccination | week 8
  To determine the effects of administration of lenalidomide combined with CD40L expressing and IL-2 secreting B-CLL cells on overall disease burden and the side population of tumor cells.
Number of patients with a tumor response post vaccination | 4 weeks
  To determine the effects of administration of lenalidomide combined with CD40L expressing and IL-2 secreting B-CLL cells on overall disease burden.
Number of patients with a tumor response post vaccination | 8 weeks
  To determine the effects of administration of lenalidomide combined with CD40L expressing and IL-2 secreting B-CLL cells on overall disease burden.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Mims, MD, Principal Investigator — Baylor College of Medicine; Malcolm Brenner, MB, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States